CLINICAL TRIAL: NCT00330564
Title: A Phase 2 Study of SU011248 (Sunitinib Malate) in Von Hippel-Lindau Syndrome
Brief Title: Evaluation of Sunitinib Malate in Patients With Von Hippel-Lindau Syndrome (VHL) Who Have VHL Lesions to Follow
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0463
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Von Hippel-Lindau Syndrome; Renal Cell Carcinoma; Hemangioblastoma
Keywords: VHL Syndrome; Von Hippel-Lindau Syndrome; VHL Disease; Kidney; Retina; Brain; Spinal cord; Pancreas; Inner ear; Cysts; Tumors; Sunitinib Malate; SU011248; Sutent; VHL; Sunitinib; Renal cell carcinoma; Hemangioblastoma; Endothelium
MeSH Terms: conditions — von Hippel-Lindau Disease; Carcinoma, Renal Cell; Hemangioblastoma; Cysts; Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SU011248 (Sutent, Sunitinib Malate) (Experimental): 50 mg/day orally for 4 weeks
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: SU011248 — 50 mg/day orally for 4 weeks, no treatment for 2 weeks (6 weeks = 1 cycle).
  Other Names: Sunitinib Malate; Sutent

SUMMARY:
The goal of this clinical research study is to learn if sunitinib malate (SU011248) can help to control VHL. The safety of this drug will also be studied.

Primary objectives:

* Evaluate safety of treatment with SU011248/sunitinib malate (50 mg daily dose for 4 weeks, then 2 weeks off) for 6 months in patients with Von Hippel-Lindau Syndrome (VHL) who have a measurable lesion undergoing surveillance

Secondary objectives:

* Evaluate efficacy of treatment with SU011248/sunitinib malate (50 mg daily dose for 4 weeks, then 2 weeks off) for 6 months in patients with VHL who have a measurable lesion undergoing surveillance

Correlative objectives:

* Evaluate quality of life of SU011248/sunitinib malate therapy in VHL patients
* Evaluate peripheral blood lymphocyte receptor phosphorylation in VHL patients taking SU011248/sunitinib malate (optional procedure)
* Correlate results of dynamic contrast-enhanced and diffusion weighted MRI and dynamic contrast enhanced CT with response and explore findings suggestive of surrogates of early response (optional procedure)

DETAILED DESCRIPTION:
Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have standard scans to check the status of your disease, including computed tomography (CT) scans of the chest and abdomen (stomach area) and/or a magnetic resonance imaging (MRI) scan of the spine, if you have lesions in these areas. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart) and an echocardiogram or MUGA scan (echocardiogram/MUGA scan - a test to determine how well your heart is functioning by measuring its ability to pump blood). If the doctors know or suspect that VHL is affecting your eyes you will have an eye exam performed.

Your complete medical history will be recorded and you will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight. You will be asked about any medications or treatments you are currently taking. Blood (about 2 teaspoons) will be drawn for routine tests. You will also be asked about your ability to perform daily activities. Women who are able to have children must have a negative blood pregnancy test.

You will be asked to complete 2 questionnaires that ask about your quality of life and your level of fatigue. It will take about 20 minutes to complete both questionnaires. The same questionnaires will then be completed 4-6 weeks later, and again at the end of treatment.

If you are found to be eligible to take part in this study, you will take sunitinib malate once a day, either with or without food. You will take the drug for 4 weeks in a row followed by 2 weeks of rest with no study drug. These 6 weeks are called a study "cycle".

Before beginning each new cycle, you will have a physical exam and your complete medical history will be recorded. Blood (about 1 teaspoon) will be drawn for routine tests. You will be asked about any drugs you have taken and any side effects you may have experienced. You will also be asked about your ability to perform daily activities.

At the end of Cycles 2 and 4, you will have CT or MRI scans to evaluate the status of your disease and eye exams may be repeated for those with known lesions on their eye(s).

You may receive treatment on this study for 24 weeks. However if you are showing benefit from the study drug, you may continue on study for an additional 24 weeks. (maximum total of 48 weeks) You will be taken off study if the disease gets worse or if intolerable side effects occur.

Once you stop treatment, you will have an end-of-study visit. At this visit, you will have a physical exam and blood (about 1 teaspoon) will be drawn for routine tests. You will be asked about any medications you have taken and any side effects you may have experienced. You will have CT or MRI scans to evaluate the status of your disease, as well as an eye exam if your eyes are affected by your disease. If you have completed at least 1 cycle of treatment on this study, and have had imaging scans in the past 28 days, you will skip the end of study evaluation and return for the 48 week follow-up visit.

You will have a follow-up visit about 48 weeks after your date of enrollment on this study. At this visit, you will have a physical exam and blood (about 1 teaspoon) will be drawn for routine tests. You will be asked about any medications you have taken and any side effects you may have experienced. You will have CT or MRI scans to evaluate the status of your disease. If your eyes are being affected by the disease, you will have a follow-up eye exam.

Once you complete the 48 week follow-up visit, you are considered off-study.

This is an investigational study. Sunitinib malate has been authorized by the FDA for research purposes only. About 28 patients will take part in this clinical research study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have genetically confirmed Von Hippel-Lindau (VHL) disease.
* At least one measurable VHL-related lesion, which is undergoing surveillance, and patient is not at immediate risk of needing intervention for this or other lesions. Biopsy is not required given the known natural history in the setting of a positive genetic test. (1) Renal: solid mass suspicious for Renal Cell Carcinoma (RCC) >/= 1 cm or cystic mass >/= 1 cm; (2) Pancreas: Solid mass >/= 1cm & < 3cm suspicious for neuroendocrine tumor; (3) Brain: asymptomatic hemangioblastoma > 5mm; (4) Spine: asymptomatic hemangioblastoma, > 1cm; (5) Eye: asymptomatic peripapillary and/or macular hemangioblastoma, any size.
* Allowable prior therapy: (1) Patients having undergone prior therapy for VHL lesions may enroll as long as other criteria are met. Previously radiated lesions may not be considered as target lesions unless they demonstrate unequivocal evidence of growth; (2) Major surgery, chemotherapy or radiation therapy completed >4 weeks prior to starting the study treatment.
* Age >/= 18 years. Because no dosing or adverse event data are currently available on the use of SU011248/sunitinib malate in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2
* Patients must have normal organ and marrow function as defined: (1) serum aspartate transaminase ([AST]; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase ([ALT]; serum glutamic pyruvic transaminase [SGPT]) </= 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT</= 5 x ULN if liver function abnormalities are due to underlying malignancy; (2) Total serum bilirubin </=1.5 x ULN; (3) Absolute neutrophil count (ANC) >/= 1500mcL; (4) Platelets >/= 100,000 mcL; (5) Hemoglobin >/= 9.0 g/dL; (6) Serum creatinine < 1.5 x UL.
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of SU011248/sunitinib malate as listed below will be determined following review of their case by the Principal Investigators. If possible, efforts will be made to switch motivated patients to other medications, otherwise patients will be excluded: (1) Ketoconazole, (2) Theophylline, (3) Phenobarbital, (4) Coumadin at therapeutic doses (low dose Coumadin up to 2 mg po daily for thromboprophylaxis is allowed).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with any metastatic disease of any kind.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SU011248/sunitinib malate.
* National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 3 hemorrhage within 4 weeks of starting the study treatment.
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening Computer tomography (CT) or Magnetic Resonance Imaging (MRI) scan.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade >/= 2.
* Prolonged QTc interval on baseline electrocardiogram (ECG or EKG)>470ms.
* Hypertension that cannot be controlled by medications (>140/90 mm Hg despite optimal medical therapy).
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because SU011248/sunitinib malate has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SU011248/sunitinib malate, breastfeeding should be discontinued if the mother is treated with SU011248/sunitinib malate.
* Known HIV-positive patients taking combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with SU011248/sunitinib malate. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Jonasch E, McCutcheon IE, Waguespack SG, Wen S, Davis DW, Smith LA, Tannir NM, Gombos DS, Fuller GN, Matin SF. Pilot trial of sunitinib therapy in patients with von Hippel-Lindau disease. Ann Oncol. 2011 Dec;22(12):2661-2666. doi: 10.1093/annonc/mdr011. PMID 22105611
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 5/19/2006 to 3/17/2010. Participants recruited from routine appointments at a Comprehensive Cancer Center.
Pre-assignment Details: Study terminated early due to slow accrual.
Period: Overall Study
Arm/Group | SU011248 (Sutent, Sunitinib Malate)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SU011248 (Sutent, Sunitinib Malate)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: participants] | 36 [22 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Secondary Outcome: Number of VHL Lesion Complete + Partial Responses
Description: Response of VHL lesions (number) evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) of Complete Response (CR): Disappearance of all target lesions, and Partial Response (PR): At least a 30% decrease in the sum of longest diameter (LD) of target lesions, reference baseline sum LD. Progressive Disease (PD): 20% increase in LD sum and Stable Disease (SD): Insufficient shrinkage to qualify for PR nor increase to qualify for PD. Degree and timing of response in affected organs evaluated in order to determine organ specific kinetics of therapy.
Time Frame: Baseline to 12 months (evaluations at 6 and 12 months)
Population: Secondary end point of efficacy showed response of renal cell carcinomas, which responded better to sunitinib therapy than other VHL related lesions using RECIST measure.
Measure: Number; unit: VHL lesion
Units Other Than Participants: renal cell carcinoma lesions
Arm/Group | SU011248 (Sutent, Sunitinib Malate)
Number analyzed (Participants) | 15
Number analyzed (renal cell carcinoma lesions) | 18
VHL lesion
  CR | 0
  PR | 6

2. Primary Outcome: Safety of Sunitinib Administration in Participants With Von Hippel-Lindau Syndrome (VHL)
Description: Safety evaluation = Number of participants with treatment terminating toxicity using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 3.0. Early stopping rules applied when treatment terminating toxicity occurred in the first 6 week cycle. Recurring grade 3 toxicity requires dose reduction, with no more than 2 dose reductions permitted. If no improvement after 4 weeks, patient is taken off drug and off study, and the event recorded as treatment terminating toxicity.
Time Frame: 12 weeks
Population: Intent to treat once the first dose was taken.
Measure: Number; unit: participants
Arm/Group | SU011248 (Sutent, Sunitinib Malate)
Number analyzed (Participants) | 15
participants | 15

ADVERSE EVENTS:
Time Frame: 3 years, 8 months
Arm/Group | SU011248 (Sutent, Sunitinib Malate)
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SU011248 (Sutent, Sunitinib Malate) (N=15)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
fatigue (General disorders) | 5 (5)
hand foot syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
hypertension (Cardiac disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations include the conclusion of the study before maximum enrollment and the use of archival tissue that was not related to the participants in the clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No